CLINICAL TRIAL: NCT03718767
Title: Phase II Trial Evaluating Nivolumab In Patients With IDH-Mutant Gliomas With And Without Hypermutator Phenotype
Brief Title: Nivolumab in Patients With IDH-Mutant Gliomas With and Without Hypermutator Phenotype
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Jing Wu, M.D., Principal Investigator, National Cancer Institute (NCI)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 190006; 19-C-0006
Record Dates: First submitted 2018-10-23; First posted 2018-10-24 (Actual); Results first posted 2025-11-24 (Actual); Last update posted 2025-11-24 (Actual); Status verified 2025-11

CONDITIONS: Glioma; Glioblastoma; High Grade Glioma; Low Grade Glioma; Malignant Glioma
Keywords: PD 1 Pathway; High Tumor Mutational Load; Immune Checkpoint; Quality of Life
MeSH Terms: conditions — Glioma; Glioblastoma | interventions — Nivolumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Arm1/Nivolumab (Experimental): Intravenous (IV) nivolumab
  Interventions: Drug: Nivolumab

INTERVENTIONS:
Drug: Nivolumab — Intravenous (IV) Nivolumab
  Other Names: Opdivo

SUMMARY:
Background:

Gliomas are the most common malignant brain tumors. Some have certain changes (mutations) in the genes isocitrate dehydrogenase 1 (IDH1) or isocitrate dehydrogenase 2 (IDH2). If there are a high number of mutations in a tumor, it is called hypermutator phenotype (HMP). The drug nivolumab helps the immune system fight cancer. Researchers think it can be more effective in patients with IDH1 or IDH2 mutated gliomas with HMP. They will test gliomas with and without HMP.

Objectives:

To see if nivolumab stops tumor growth and prolongs the time that the tumor is controlled.

Eligibility:

Adults 18 years or older with IDH1 or IDH2 mutated gliomas

Design:

Participants will be screened with:

Medical history

Physical exam

Heart, blood, and pregnancy tests

Review of symptoms and activity levels

Brain magnetic resonance imaging (MRI). Participants will lie in a cylinder that takes pictures in a strong magnetic field.

Tumor samples

Participants will get the study drug in 4-week cycles. They will get it through a small plastic tube in a vein (intravenous [IV]) on days 1 and 15 of cycles 1-4. For cycles 5-16, they will get it just on day 1.

On days 1 and 15 of each cycle, participants will repeat some or all screening tests.

After cycle 16, participants will have 3 follow-up visits over 100 days. They will answer health questions, have physical and neurological exams, and have blood tests. They may have a brain MRI.

Participants whose disease did not get worse but who finished the study drug within 1 year of treatment may have imaging studies every 8 weeks for up to 1 year.

Participants will be called or emailed every 6 months with questions about their health.

DETAILED DESCRIPTION:
BACKGROUND:

* Glioma is the most common malignant brain tumor. Genes coding for isocitrate dehydrogenases 1and 2 (IDH1 and IDH2), metabolic enzymes, are frequently mutated in gliomas, particularly lower-grade gliomas (LGGs). IDH1/2 mutation causes a unique tumor biology, including the accumulation of 2-hydroxyglutarate (2-HG), an oncometabolite, which in turn causes genomic hypermethylation and tumorigenesis.
* IDH-mutant LGGs undergo a slow but unremitting progression to higher grade transformation (HT) and eventually become high grade gliomas (HGGs) with a significant increase in the number of somatic mutations. A subset of patients with transformed HGGs develop a hypermutator phenotype (HMP), possibly related, but not limited, to previous treatment with alkylating agents and radiotherapy. The mechanisms of this clinical phenomenon are not fully understood, and no effective treatments are available for the HMP HGGs.
* High tumor mutation burden (TMB) is a characteristic finding in many of the transformed tumors. Furthermore, this increased mutation burden, with commensurate increase in neoantigen expression, may be correlated with a better response to immune checkpoint inhibitor (ICPIs) treatment.
* Nivolumab is a monoclonal antibody that binds to the programmed cell death protein 1 (PD1) receptor and blocks its interaction with programmed death-ligand 1 (PD L1) and PD L2 and subsequently releasing PD 1 pathway mediated inhibition of the immune response, including antitumor immune response.
* The United States (US) Food and Drug Administration granted approval to nivolumab for the treatment of unresectable or metastatic melanoma, advanced non-small cell lung cancer, renal cell carcinoma, Hodgkin's lymphoma, recurrent or metastatic squamous cell carcinoma of the head and neck, locally advanced or metastatic urothelial carcinoma, microsatellite instability-high or mismatched repair deficient metastatic colorectal cancer and hepatocellular carcinoma.
* The first randomized clinical trial in glioblastoma with nivolumab (CheckMate-143) was completed in early 2017. Unfortunately, the study didn't meet its primary endpoint of improved overall survival over bevacizumab monotherapy. The objective response rate (ORR) was lower in nivolumab arm than bevacizumab arm. However, the response with nivolumab was more durable. The safety profile of nivolumab was very consistent with what has been observed in other tumor types.

OBJECTIVE:

-To determine the 6-month progression free survival rate in IDH-mutant gliomas patients with and without HMP in responses to nivolumab treatment.

ELIGIBILITY:

* Patients with diffuse glioma, confirmed by National Cancer Institute (NCI) Laboratory of Pathology
* Age greater than or equal to 18 years
* Karnofsky Performance Scale (KPS) greater than or equal to 60%
* IDH 1 or IDH 2 mutation confirmed by deoxyribonucleic acid (DNA) sequencing
* Patients must have TMB status performed at National Institutes of Health (NIH)
* Tumor tissue or slides should be available for molecular and immune profiling

DESIGN:

* This study is an open label phase II clinical trial of the immune checkpoint inhibitor, nivolumab, in patients with HMP and non-hypermutated phenotype (NHMP) IDH-mutant gliomas.
* Patients with HMP and NHMP will receive nivolumab at a standard dose of 240 mg intravenously every 2 weeks for cycles 1-2, then doses of 480 mg every 4 weeks for cycles 3-16. A maximum of 20 treatments will be given (16 cycles).
* A maximum of 29 patients with IDH-mutant glioma with HMP (Cohort 1) and 30 patients with NHMP (Cohort 2) will be evaluated.
* A Simon's optimal two-stage design will be used to conduct the HMP arm and the NHMP arm independently. For the HMP cohort, in stage I, a total number of 10 patients are accrued. If 9 or more patients progress by 6 months, the cohort will be terminated early; otherwise, additional 19 patients will be accrued in stage II, resulting in a total sample size of 29. Among these 29 patients, if 6 or more patients are progression-free at 6 months, we will claim that the treatment is promising for patients with HMP IDH-mutant gliomas. For NHMP cohort, in stage I, a total number of 15 patients are accrued. If 3 or more patients are progression-free at 6 months, the cohort will move to stage II and an additional 15 patients will be accrued in stage II, resulting in a total sample size of 30. Among these 30 patients, if 10 or more patients are progression-free at 6 months, we will claim that the treatment is promising for patients with NHMP IDH-mutant gliomas.

ELIGIBILITY:
* INCLUSION CRITERIA:
* Patients must have recurrent diffuse glioma (histologically confirmed by National Institutes of Health (NIH) Laboratory of Pathology) with isocitrate dehydrogenase 1 (IDH1) or isocitrate dehydrogenase 2 (IDH2) mutation (confirmed by deoxyribonucleic acid (DNA) sequencing, Foundation One is preferable for confirmation of mutation, but not necessary).
* Patients must have tumor specific mutation burden (number of somatic mutations per exome) tested at NIH: Must have either result of tumor mutation burden from the most recent surgical tumor sample or must provide adequate genomic materials of the sample for tumor testing. The tumor tissue (e.g., block or 15 unstained slides) must be available for molecular and immune profiling. Fresh or frozen tumor sample will be used if available, but not mandatory.
* Age greater than or equal to 18 years. Because no dosing or adverse event data are currently available on the use of nivolumab in patients <18 years of age, children are excluded from this study but will be eligible for future pediatric trials.
* Patient must be able to tolerate a magnetic resonance imaging (MRI) study with intravenous gadolinium contrast.
* Karnofsky greater than or equal to 60%
* Patients must have adequate organ and marrow function as defined below:

  * Absolute neutrophil count greater than or equal to 1,500/mcL
  * Platelet Count greater than or equal to 100,000/MCL
  * Hemoglobin greater than 9.0 g/dL (may be transfused to achieve this level)
  * Blood Urea Nitrogen (BUN) less than or equal to 30 mg/dL and
  * Serum creatinine less than or equal to 1.7 mg/dL
  * Total bilirubin (except patients with Gilbert's Syndrome, who are eligible for the study but exempt from the total bilirubin eligibility criterion) less than or equal to 2.0 mg/dL
  * Alanine aminotransferase (ALT) and aspartate aminotransaminase (AST) less than or equal to 2.5x institutional upper limit of normal.
* The effects of nivolumab on the developing human fetus are unknown. For this reason, women of child-bearing potential must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation and up to 5 months (women). Should a woman become pregnant or suspect she is pregnant while she is participating in this study, she should inform her treating physician immediately.
* The patient must be able to understand and be willing to sign a written informed consent document.

EXCLUSION CRITERIA:

* Patients who are receiving any other investigational agents.
* Patients who have a history of receiving immune therapy.
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to nivolumab.
* History of severe hypersensitivity reaction to any monoclonal antibody.
* Prior invasive malignancy (except non-melanomatous skin cancer) unless disease free for a minimum of 3 years prior to initiation of study therapy.
* Patients with active autoimmune disease or history of autoimmune disease that might recur, which may affect vital organ function or require immune suppressive treatment including systemic corticosteroids. These include but are not limited to patients with a history of immune related neurologic disease, multiple sclerosis, autoimmune (demyelinating) neuropathy, Guillain-Barre syndrome or Chronic Inflammatory Demyelinating Polyneuropathy (CIDP), myasthenia gravis; systemic autoimmune disease such as Systemic Lupus Erythematosus (SLE), connective tissue diseases, scleroderma, inflammatory bowel disease (IBD), Crohn's, ulcerative colitis, hepatitis; and patients with a history of toxic epidermal necrolysis (TEN), Stevens-Johnson syndrome, or phospholipid syndrome. Such diseases should be excluded because of the risk of recurrence or exacerbation of disease.

  --Of note, patients with vitiligo, endocrine deficiencies including thyroiditis managed with replacement hormones including physiologic corticosteroids are eligible. Patients with rheumatoid arthritis and other arthropathies, Sjogren's syndrome and psoriasis controlled with topical medication and patients with positive serology, such as antinuclear antibodies (ANA), anti-thyroid antibodies should be evaluated for the presence of target organ involvement and potential need for systemic treatment but should otherwise be eligible.
* The patient must not be currently on a corticosteroid dose greater than dexamethasone 1 mg per day or its equivalent.
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations (within timeframes identified in the bullets below) that would limit compliance with study requirements.
* Known human immunodeficiency virus (HIV)-positive or acquired immune deficiency syndrome (AIDS) based upon current Centers for Disease Control and Prevention (CDC) definition; note, however, that HIV testing is not required for entry into this protocol. The need to exclude patients with AIDS is based on the lack of information regarding the safety of nivolumab in patients with active HIV infection
* Pregnant women are excluded from this study because nivolumab's potential for teratogenic or abortifacient effects is unknown. Because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with nivolumab, breastfeeding should be discontinued if the mother is treated with nivolumab.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2019-03-27 (Actual); Primary Completion 2024-11-05 (Actual); Study Completion 2026-11-30 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Jing Wu, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
Biomedical Translational Research Information System (BTRIS): All individual participant data (IPD) recorded in the medical record will be shared with intramural investigators upon request. The database of Genotypes and Phenotypes (dbGaP): All large-scale genomic sequencing data will be shared with subscribers to dbGaP.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Biomedical Translational Research Information System (BTRIS): Clinical data available during the study and indefinitely. The database of Genotypes and Phenotypes (dbGaP): Genomic data are available once genomic data are uploaded per protocol Genomic Data Sharing (GDS) plan for as long as database is active.
Access Criteria: Biomedical Translational Research Information System (BTRIS): Clinical data will be made available via subscription to BTRIS and with the permission of the study principal investigator (PI). The database of Genotypes and Phenotypes (dbGaP): Genomic data are made available via dbGaP through requests to the data custodians.

REFERENCES:
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2019-C-0006.html

RESULTS

PARTICIPANT FLOW:
Groups:
- Cohort 1/Hypermutated Phenotype (HMP): Isocitrate dehydrogenase (IDH) - mutant gliomas participants with hypermutated phenotype (HMP). Participants received Nivolumab 240mg every (q)2 weeks in Cycle 1 - Cycle 2 and then 480mg q4 weeks in Cycle 3-Cycle 16.
- Cohort 2/Non-hypermutated Phenotype (NHMP).: Isocitrate dehydrogenase (IDH) - mutant gliomas participants with non-hypermutated phenotype (NHMP). Participants received Nivolumab 240mg every (q)2 weeks in Cycle 1 - Cycle 2 and then 480mg q4 weeks in Cycle 3-Cycle 16.
- Enrolled But Not Treated: Participants were enrolled, not assigned to Cohorts/Arms and not treated.
Period: Overall Study
Arm/Group | Cohort 1/Hypermutated Phenotype (HMP) | Cohort 2/Non-hypermutated Phenotype (NHMP). | Enrolled But Not Treated
Started | 8 | 30 | 24
Completed | 8 | 30 | 0
Not Completed | 0 | 0 | 24
Not completed — Declined to participate (before treatment started) | 0 | 0 | 7
Not completed — Ineligible | 0 | 0 | 17

BASELINE CHARACTERISTICS:
Population: Baseline characteristics is reported for participants enrolled but not treated.
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort 1/Hypermutated Phenotype (HMP) | Cohort 2/Non-hypermutated Phenotype (NHMP). | Enrolled But Not Treated | Total
Number analyzed (Participants) | 8 | 30 | 24 | 62
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 8 | 28 | 24 | 60
  >=65 years | 0 | 2 | 0 | 2
Age, Continuous [Mean (Standard Deviation); unit: years] | 44.38 (11.7) | 45.27 (11.68) | 40.5 (10.19) | 43.31 (11.17)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 10 | 6 | 21
  Male | 3 | 20 | 18 | 41
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Ethnicity: Hispanic or Latino | 8 | 4 | 1 | 13
  Ethnicity: Not Hispanic or Latino | 0 | 26 | 23 | 49
  Ethnicity: Unknown or Not Reported | 0 | 0 | 0 | 0
  Race: American Indian or Alaska Native | 0 | 0 | 0 | 0
  Race: Asian | 0 | 5 | 0 | 5
  Race: Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Race: Black or African American | 0 | 1 | 2 | 3
  Race: White | 8 | 21 | 21 | 50
  Race: More than one race | 0 | 0 | 1 | 1
  Race: Unknown or Not Reported | 0 | 2 | 00 | 2
  Race: Other | 0 | 1 | 0 | 1
Region of Enrollment [Number; unit: participants]
  United States | 8 | 30 | 24 | 62

OUTCOME MEASURES:

1. Primary Outcome: Median Progression Free Survival (PFS) Rate at 6 Months
Description: PFS is defined from the day of study entry until imaging is confirmed to show disease progression or death, whichever occurs first. Disease progression was assessed by the Immunotherapy Response Assessment neuro-oncology Criteria. Disease progression is >25% increase in sum of the products of perpendicular diameters of enhancing lesions; any new enhancing measurable lesion that exceeds a 25% increase in cross-sectional area; clear clinical deterioration not attributable to other causes apart from the tumor and/or failure to return for evaluation due to death or deteriorating condition. PFS was analyzed by the Kaplan-Meier method and is reported with a 95% confidence interval.
Time Frame: 6 months
Population: 38/62 participants are reported because 7 declined to participate (before treatment started) and 17 were ineligible.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Cohort 1/Hypermutated Phenotype (HMP) | Cohort 2/Non-hypermutated Phenotype (NHMP).
Number analyzed (Participants) | 8 | 30
Percentage of participants | 25.0 [7.5 to 83.0] | 40.0 [25.8 to 62.0]

2. Secondary Outcome: Mean Symptom Interference Score Per Treatment Cycle Using the MD Anderson Symptom Inventory-Brain Tumor Module (MDSAI-BT)
Description: Participant reported outcome measures using self-reported symptom interference with daily activities using the MD Anderson Symptom Inventory-Brain Tumor Module (MDSAI-BT). The MDSAI-BT 5-minute questionnaire uses an 11-point scale (0-10) to rate symptoms interference in the last 24 hours of a participant's life related to mood, work Inside and outside the home), relations with other people, walking and enjoyment of life. 0 = symptom not present and 10 = as bad as you can imagine. Higher score indicates more interference. Per protocol, MDSAIs are performed with imaging. If no imaging, no MDASI.
Time Frame: Baseline and Cycles 2, 4, 6, 8, 10, 12, 14, and 16 (approximately 32 weeks +/- 3 days).
Population: 38/62 participants were reported because 7 declined to participate (before treatment started) and 17 were ineligible. Reasons data not reported in Cycles: participants came off treatment due to disease progression or toxicity, refused further treatment, did not complete the questionnaire, did extra MDASI because of short-interval imaging, refused to complete MDASI (no computer), data collected but not captured in database for a participant, and MDSAI not done related to outside hospitalization.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Cohort 1/Hypermutated Phenotype (HMP) | Cohort 2/Non-hypermutated Phenotype (NHMP).
Number analyzed (Participants) | 8 | 30
score on a scale
  Baseline | 3.96 (2.96) | 2.06 (2.80)
  Cycle 2: number analyzed (Participants) | 7 | 25
  Cycle 2 | 3.21 (2.67) | 2.30 (2.35)
  Cycle 4: number analyzed (Participants) | 4 | 15
  Cycle 4 | 2.33 (1.99) | 2.19 (2.07)
  Cycle 6: number analyzed (Participants) | 2 | 9
  Cycle 6 | 2.42 (3.42) | 2.41 (2.06)
  Cycle 8: number analyzed (Participants) | 2 | 8
  Cycle 8 | 3.00 (4.00) | 2.46 (2.03)
  Cycle 10: number analyzed (Participants) | 2 | 7
  Cycle 10 | 4.17 (5.42) | 1.45 (1.43)
  Cycle 12: number analyzed (Participants) | 2 | 8
  Cycle 12 | 4.25 (6.01) | 1.00 (1.28)
  Cycle 14: number analyzed (Participants) | 2 | 6
  Cycle 14 | 4.83 (6.36) | 1.17 (1.59)
  Cycle 16: number analyzed (Participants) | 0 | 5
  Cycle 16 |  | 0.57 (1.27)

3. Secondary Outcome: Mean Symptom Severity Score Per Treatment Cycle Using the MD Anderson Symptom Inventory-Brain Tumor Module (MDSAI-BT)
Description: Participant reported outcome measures using self-reported symptom severity with daily activities (e.g., work) using the MD Anderson Symptom Inventory-Brain Tumor Module (MDSAI-BT) are reported for each treatment cycle. The MDSAI-BT 5-minute questionnaire uses an 11-point Likert scale (0-10). 0 = symptom not present and 10 = as bad as you can imagine. Higher score indicates worse severity. Per protocol, MDSAIs are performed with imaging. If no imaging, no MDASI.
Time Frame: Baseline and Cycles 2, 4, 6, 8, 10, 12, 14, and 16 (approximately 32 weeks +/- 3 days).
Population: 38/62 participants were reported because 7 declined to participate (before treatment started) and 17 were ineligible.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Cohort 1/Hypermutated Phenotype (HMP) | Cohort 2/Non-hypermutated Phenotype (NHMP).
Number analyzed (Participants) | 8 | 30
score on a scale
  Baseline | 3.16 (2.78) | 4.16 (1.56)
  Cycle 2: number analyzed (Participants) | 7 | 25
  Cycle 2 | 2.16 (1.77) | 1.48 (1.29)
  Cycle 4: number analyzed (Participants) | 4 | 15
  Cycle 4 | 1.61 (1.31) | 1.50 (1.23)
  Cycle 6: number analyzed (Participants) | 2 | 9
  Cycle 6 | 2.00 (2.57) | 1.26 (1.12)
  Cycle 8: number analyzed (Participants) | 2 | 8
  Cycle 8 | 1.91 (2.57) | 1.20 (1.25)
  Cycle 10: number analyzed (Participants) | 2 | 7
  Cycle 10 | 2.07 (2.80) | 0.82 (0.70)
  Cycle 12: number analyzed (Participants) | 2 | 8
  Cycle 12 | 2.70 (3.70) | 0.97 (0.97)
  Cycle 14: number analyzed (Participants) | 2 | 6
  Cycle 14 | 2.41 (3.34) | 0.74 (0.51)
  Cycle 16: number analyzed (Participants) | 0 | 5
  Cycle 16 |  | 0.72 (0.81)

4. Secondary Outcome: Overall Survival
Description: OS is defined as the time from treatment initiation to the time of death.
Time Frame: Until the death of the last surviving participant, a median of 7.4 months in Cohort 1 and a median of 31.6 months in Cohort 2.
Population: 38/62 participants are reported because 7 declined to participate (before treatment started) and 17 were ineligible.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Cohort 1/Hypermutated Phenotype (HMP) | Cohort 2/Non-hypermutated Phenotype (NHMP).
Number analyzed (Participants) | 8 | 30
Months | 7.4 [4.7 to NA] — The upper confidence interval is not reported because participants were not evaluable. | 31.6 [10.2 to NA] — The upper confidence interval is not reported because participants were not evaluable.

5. Secondary Outcome: Tumor Mutation Burden
Description: Tumor mutation Burden is measured using whole exome sequencing.
Time Frame: During the screening period (14 days prior to study therapy)
Population: 38/62 participants were reported because 7 declined to participate (before treatment started) and 17 were ineligible.
Measure: Mean (Standard Deviation); unit: mutation/Mb
Arm/Group | Cohort 1/Hypermutated Phenotype (HMP) | Cohort 2/Non-hypermutated Phenotype (NHMP).
Number analyzed (Participants) | 8 | 30
mutation/Mb | 76.39 (78.54) | 1.28 (0.61)
Statistical Analysis 1: Comparison: Cohort 1/Hypermutated Phenotype (HMP); Test type: Other; p = 0.623, Regression, Cox; Hazard Ratio (HR) = 1
Statistical Analysis 2: Comparison: Cohort 2/Non-hypermutated Phenotype (NHMP); Test type: Other; p = 0.073, Regression, Cox; Hazard Ratio (HR) = 1.73

6. Secondary Outcome: Proportion of Participants Rating Symptoms 5 or Greater (on a 0-10 Scale) Using the MD Anderson Symptom Inventory-Brain Tumor Module (MDSAI-BT)
Description: The proportion of participants rating symptoms 5 or greater (on a 0-10 scale) was assessed using the MD Anderson Symptom Inventory-Brain Tumor Module (MDSAI-BT). The MD Anderson Symptom Inventory-Brain Tumor Module (MDSAI-BT) 5-minute questionnaire uses an 11-point Likert scale (0-10) to measure symptoms reported by the participant. 0 = symptom not present and 10 = as bad as you can imagine. Higher score indicates worse severity.
Time Frame: Baseline and Cycles 2, 4, 6, 8, 10, 12, 14, and 16 (approximately 32 weeks +/- 3 days).
Population: 38/62 participants were reported because 7 declined to participate (before treatment started) and 17 were ineligible.
Measure: Number; unit: proportion of participants
Groups:
- Cohort 1/Hypermutated Phenotype (HMP) - Baseline; Cohort 1/Hypermutated Phenotype (HMP) - Cycle 2; Cohort 1/Hypermutated Phenotype (HMP) - Cycle 4; Cohort 1/Hypermutated Phenotype (HMP) - Cycle 6; Cohort 1/Hypermutated Phenotype (HMP) - Cycle 8; Cohort 1/Hypermutated Phenotype (HMP) - Cycle 10; Cohort 1/Hypermutated Phenotype (HMP) - Cycle 12; Cohort 1/Hypermutated Phenotype (HMP) - Cycle 16: Isocitrate dehydrogenase (IDH) - mutant gliomas participants with hypermutated phenotype (HMP). Participants received Nivolumab 240mg every (q)2 weeks in Cycle 1 - Cycle 2 and then 480mg q4 weeks in Cycle 3-Cycle 16.
- Cohort 1/Hypermutated Phenotype (HMP) - Cycle 14: Isocitrate dehydrogenase (IDH) - mutant gliomas participants with hypermutated phenotype (HMP). Participants received Nivolumab/dose level 1 - 240mg every (q)2 weeks in Cycle 1 - Cycle 2 and then dose level 2, 480mg q4 weeks in Cycle 3-Cycle 16.
- Cohort 2/Non-hypermutated Phenotype (NHMP) - Baseline; Cohort 2/Non-hypermutated Phenotype (NHMP) - Cycle 2; Cohort 2/Non-hypermutated Phenotype (NHMP) - Cycle 4; Cohort 2/Non-hypermutated Phenotype (NHMP) - Cycle 6; Cohort 2/Non-hypermutated Phenotype (NHMP) - Cycle 8; Cohort 2/Non-hypermutated Phenotype (NHMP) - Cycle 10; Cohort 2/Non-hypermutated Phenotype (NHMP) - Cycle 12; Cohort 2/Non-hypermutated Phenotype (NHMP) - Cycle 14; Cohort 2/Non-hypermutated Phenotype (NHMP) - Cycle 16: Isocitrate dehydrogenase (IDH) - mutant gliomas participants with non-hypermutated phenotype (NHMP). Participants received Nivolumab 240mg every (q)2 weeks in Cycle 1 - Cycle 2 and then 480mg q4 weeks in Cycle 3-Cycle 16.
Arm/Group | Cohort 1/Hypermutated Phenotype (HMP) - Baseline | Cohort 1/Hypermutated Phenotype (HMP) - Cycle 2 | Cohort 1/Hypermutated Phenotype (HMP) - Cycle 4 | Cohort 1/Hypermutated Phenotype (HMP) - Cycle 6 | Cohort 1/Hypermutated Phenotype (HMP) - Cycle 8 | Cohort 1/Hypermutated Phenotype (HMP) - Cycle 10 | Cohort 1/Hypermutated Phenotype (HMP) - Cycle 12 | Cohort 1/Hypermutated Phenotype (HMP) - Cycle 14 | Cohort 1/Hypermutated Phenotype (HMP) - Cycle 16 | Cohort 2/Non-hypermutated Phenotype (NHMP) - Baseline | Cohort 2/Non-hypermutated Phenotype (NHMP) - Cycle 2 | Cohort 2/Non-hypermutated Phenotype (NHMP) - Cycle 4 | Cohort 2/Non-hypermutated Phenotype (NHMP) - Cycle 6 | Cohort 2/Non-hypermutated Phenotype (NHMP) - Cycle 8 | Cohort 2/Non-hypermutated Phenotype (NHMP) - Cycle 10 | Cohort 2/Non-hypermutated Phenotype (NHMP) - Cycle 12 | Cohort 2/Non-hypermutated Phenotype (NHMP) - Cycle 14 | Cohort 2/Non-hypermutated Phenotype (NHMP) - Cycle 16
Number analyzed (Participants) | 8 | 7 | 4 | 2 | 2 | 2 | 2 | 2 | 0 | 30 | 25 | 15 | 9 | 8 | 7 | 8 | 6 | 5
proportion of participants
  Pain | 0.38 | 0.14 | 0.25 | 0.50 | 0.50 | 0.50 | 0.50 | 0.00 |  | 0.10 | 0.08 | 0.13 | 0.11 | 0.13 | 0.00 | 0.00 | 0.00 | 0.00
  Fatigue | 0.38 | 0.43 | 0.25 | 0.50 | 0.50 | 0.50 | 0.50 | 0.50 |  | 0.33 | 0.24 | 0.47 | 0.33 | 0.38 | 0.29 | 0.38 | 0.17 | 0.40
  Nausea | 0.25 | 0.14 | 0.00 | 0.00 | 0.50 | 0.00 | 0.00 | 0.00 |  | 0.07 | 0.00 | 0.00 | 0.00 | 0.13 | 0.00 | 0.00 | 0.00 | 0.00
  Disturbed sleep | 0.25 | 0.29 | 0.25 | 0.50 | 0.50 | 0.50 | 0.50 | 0.50 |  | 0.17 | 0.16 | 0.27 | 0.11 | 0.25 | 0.00 | 0.13 | 0.00 | 0.20
  Feeling distressed | 0.38 | 0.29 | 0.25 | 0.50 | 0.50 | 0.50 | 0.50 | 0.50 |  | 0.10 | 0.12 | 0.07 | 0.00 | 0.13 | 0.00 | 0.00 | 0.00 | 0.00
  Shortness of breath | 0.25 | 0.14 | 0.00 | 0.00 | 0.00 | 0.00 | 0.00 | 0.00 |  | 0.03 | 0.00 | 0.00 | 0.00 | 0.00 | 0.00 | 0.00 | 0.00 | 0.00
  Difficulty remembering | 0.38 | 0.14 | 0.25 | 0.50 | 0.00 | 0.00 | 0.50 | 0.50 |  | 0.20 | 0.20 | 0.33 | 0.00 | 0.13 | 0.14 | 0.25 | 0.17 | 0.20
  Lack of appetite | 0.25 | 0.00 | 0.00 | 0.00 | 0.00 | 0.00 | 0.00 | 0.00 |  | 0.07 | 0.04 | 0.00 | 0.00 | 0.00 | 0.14 | 0.00 | 0.00 | 0.00
  Feeling drowsy | 0.25 | 0.14 | 0.25 | 0.50 | 0.00 | 0.00 | 0.50 | 0.00 |  | 0.20 | 0.20 | 0.40 | 0.33 | 0.25 | 0.14 | 0.13 | 0.17 | 0.20
  Dry mouth | 0.25 | 0.14 | 0.25 | 0.50 | 0.50 | 0.50 | 0.50 | 0.50 |  | 0.10 | 0.16 | 0.13 | 0.11 | 0.13 | 0.00 | 0.00 | 0.00 | 0.00
  Feeling sad | 0.50 | 0.29 | 0.25 | 0.50 | 0.50 | 0.50 | 0.50 | 0.50 |  | 0.10 | 0.08 | 0.07 | 0.00 | 0.00 | 0.00 | 0.00 | 0.00 | 0.00
  Vomiting | 0.13 | 0.00 | 0.00 | 0.00 | 0.00 | 0.00 | 0.00 | 0.00 |  | 0.03 | 0.00 | 0.00 | 0.00 | 0.13 | 0.00 | 0.00 | 0.00 | 0.00
  Numbness/Tingling | 0.38 | 0.00 | 0.00 | 0.00 | 0.00 | 0.50 | 0.50 | 0.50 |  | 0.03 | 0.16 | 0.07 | 0.11 | 0.00 | 0.00 | 0.00 | 0.00 | 0.00
  Weakness on one side of body | 0.38 | 0.43 | 0.75 | 0.50 | 0.50 | 0.50 | 0.50 | 0.50 |  | 0.20 | 0.16 | 0.20 | 0.11 | 0.13 | 0.00 | 0.13 | 0.00 | 0.20
  Difficulty understanding | 0.25 | 0.29 | 0.25 | 0.00 | 0.00 | 0.00 | 0.00 | 0.00 |  | 0.13 | 0.08 | 0.20 | 0.00 | 0.00 | 0.00 | 0.13 | 0.00 | 0.00
  Difficulty speaking | 0.38 | 0.14 | 0.00 | 0.00 | 0.50 | 0.50 | 0.50 | 0.50 |  | 0.20 | 0.28 | 0.20 | 0.00 | 0.00 | 0.00 | 0.13 | 0.00 | 0.00
  Seizure | 0.13 | 0.00 | 0.00 | 0.00 | 0.00 | 0.00 | 0.50 | 0.50 |  | 0.07 | 0.00 | 0.00 | 0.00 | 0.00 | 0.00 | 0.00 | 0.00 | 0.00
  Difficulty concentrating | 0.25 | 0.29 | 0.25 | 0.00 | 0.00 | 0.00 | 0.50 | 0.50 |  | 0.17 | 0.20 | 0.13 | 0.22 | 0.13 | 0.00 | 0.13 | 0.00 | 0.00
  Vision | 0.13 | 0.14 | 0.00 | 0.00 | 0.00 | 0.00 | 0.00 | 0.50 |  | 0.13 | 0.16 | 0.20 | 0.33 | 0.25 | 0.14 | 0.13 | 0.17 | 0.20
  Change in appearance | 0.13 | 0.00 | 0.00 | 0.00 | 0.00 | 0.00 | 0.00 | 0.50 |  | 0.13 | 0.12 | 0.20 | 0.22 | 0.13 | 0.14 | 0.25 | 0.17 | 0.40
  Change in bowel pattern | 0.13 | 0.14 | 0.00 | 0.00 | 0.00 | 0.00 | 0.00 | 0.00 |  | 0.10 | 0.08 | 0.07 | 0.00 | 0.13 | 0.00 | 0.00 | 0.00 | 0.00
  Irritability | 0.25 | 0.14 | 0.00 | 0.50 | 0.50 | 0.00 | 0.50 | 0.50 |  | 0.10 | 0.12 | 0.07 | 0.11 | 0.00 | 0.00 | 0.00 | 0.00 | 0.00
  Rash | 0.17 | 0.00 | 0.00 | 0.00 | 0.00 | 0.00 | 0.50 | 0.00 |  | 0.04 | 0.09 | 0.07 | 0.00 | 0.00 | 0.00 | 0.00 | 0.00 | 0.00

7. Secondary Outcome: Median Percentage of Participants That Have Progressive Disease At 12 Months
Description: PFS was analyzed by the Kaplan-Meier method and is reported with a 95% confidence interval. PFS is defined from the day of study entry until imaging is confirmed to show disease progression. Disease progression was assessed by the Immunotherapy Response Assessment neuro-oncology Criteria. Disease progression is >25% increase in sum of the products of perpendicular diameters of enhancing lesions; any new enhancing measurable lesion that exceeds a 25% increase in cross-sectional area; clear clinical deterioration not attributable to other causes apart from the tumor and/or failure to return for evaluation due to death or deteriorating condition.
Time Frame: At 12 months
Population: 38/62 participants were reported because 7 declined to participate (before treatment started) and 17 were ineligible.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Cohort 1/Hypermutated Phenotype (HMP) | Cohort 2/Non-hypermutated Phenotype (NHMP).
Number analyzed (Participants) | 8 | 30
Percentage of participants | 25.0 [7.5 to 83.0] | 33.3 [20.1 to 55.3]

8. Secondary Outcome: Number of Participants Responses Received and Were Expected Using the MD Anderson Symptom Inventory-Brain Tumor Module (MDSAI-BT) Forms
Description: Here is the number of participants with IDH-mutant gliomas with and without hypermutator phenotype, responses received and were expected using the MD Anderson Symptom Inventory-Brain Tumor Module (MDSAI-BT) forms. Received MDASI-BT forms will be checked versus the timing schedule and considered as valid if they fall within ten days of the scheduled assessment window. Compliance rates will be calculated as the number of received valid forms over the number of expected forms.
Time Frame: Baseline and Cycles 2, 4, 6, 8, 10, 12, 14, and 16 (approximately 32 weeks +/- 3 days).
Population: 38/62 participants were reported because 7 declined to participate (before treatment started) and 17 were ineligible.
Measure: Count of Participants; unit: Participants
Groups:
- Cohort 1/Hypermutated Phenotype (HMP): Isocitrate dehydrogenase (IDH) - mutant gliomas participants with hypermutated phenotype (HMP). Participants received Nivolumab/ 240mg every (q)2 weeks in Cycle 1 - Cycle 2 and then 480mg q4 weeks in Cycle 3-Cycle 16.
- Cohort 2/Non-hypermutated Phenotype (NHMP): Isocitrate dehydrogenase (IDH) - mutant gliomas participants with non-hypermutated phenotype (NHMP). Participants received Nivolumab/dose level 1 - 240mg every (q)2 weeks in Cycle 1 - Cycle 2 and then dose level 2, 480mg q4 weeks in Cycle 3-Cycle 16.
Arm/Group | Cohort 1/Hypermutated Phenotype (HMP) | Cohort 2/Non-hypermutated Phenotype (NHMP)
Number analyzed (Participants) | 8 | 30
Participants
  Expected at baseline | 8 | 30
  Received at baseline | 8 | 30
  Expected at Cycle 2 | 7 | 27
  Received at Cycle 2 | 7 | 25
  Expected at Cycle 4 | 4 | 16
  Received at Cycle 4 | 4 | 15
  Expected at Cycle 6 | 2 | 11
  Received at Cycle 6 | 2 | 9
  Expected at Cycle 8 | 2 | 9
  Received at Cycle 8 | 2 | 8
  Expected at Cycle 10 | 2 | 8
  Received at Cycle 10 | 2 | 7
  Expected at Cycle 12 | 2 | 8
  Received at Cycle 12 | 2 | 8
  Expected at Cycle 14 | 2 | 7
  Received at Cycle 14 | 2 | 6
  Expected at Cycle 16 | 2 | 7
  Received at Cycle 16 | 0 | 5

9. Other Pre Specified Outcome: Number of Participants With Serious and/or Non-serious Adverse Events Assessed by the Common Terminology Criteria for Adverse Events (CTCAE v5.0)
Description: Here is the number of participants with serious and/or non-serious adverse events assessed by the Common Terminology Criteria for Adverse Events (CTCAE v5.0). A non-serious adverse event is any untoward medical occurrence. A serious adverse event is an adverse event or suspected adverse reaction that results in death, a life-threatening adverse drug experience, hospitalization, disruption of the ability to conduct normal life functions, congenital anomaly/birth defect or important medical events that jeopardize the patient or subject and may require medical or surgical intervention to prevent one of the previous outcomes mentioned.
Time Frame: From the first study intervention, Study Day 1 of Cycle 1 through 30 days after the study agent (s) was/were administered, up to 17 months
Population: 38/62 participants were reported because 7 declined to participate (before treatment started) and 17 were ineligible.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1/Hypermutated Phenotype (HMP) | Cohort 2/Non-hypermutated Phenotype (NHMP).
Number analyzed (Participants) | 8 | 30
Participants | 7 | 26

ADVERSE EVENTS:
Time Frame: All-Cause Mortality was monitored/assessed up to a median of 7.4 months in cohort 1 and a median of 31.6 months in cohort 2. Adverse Events (AEs) were only collected from beginning of study participation to one month post study participation, a maximum of 17 months.
Description: 38/62 participants are reported because 7 declined to participate (before treatment started) &17 were ineligible.
Arm/Group | Cohort 1/Hypermutated Phenotype (HMP) | Cohort 2/Non-hypermutated Phenotype (NHMP).
All-Cause Mortality (participants affected / at risk) | 6/8 | 16/30
Serious Adverse Events (participants affected / at risk) | 3/8 | 11/30
Other Adverse Events (participants affected / at risk) | 7/8 | 26/30
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1/Hypermutated Phenotype (HMP) (N=8) | Cohort 2/Non-hypermutated Phenotype (NHMP). (N=30)
Confusion (Psychiatric disorders) | 1 (1) | 1 (1)
Disease progression (General disorders) | 1 (1) | 2 (2)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1)
Edema cerebral (Nervous system disorders) | 0 (0) | 2 (2)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Fatigue (General disorders) | 0 (0) | 1 (1)
Gastrointestinal disorders - Other, specify: Immune-mediated colitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
General disorders and administration site conditions - Other, specify: Disease Progression (General disorders) | 0 (0) | 1 (1)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 1 (1)
Intracranial hemorrhage (Nervous system disorders) | 0 (0) | 2 (2)
Lung infection (Infections and infestations) | 0 (0) | 1 (1)
Nervous system disorders - Other, specify: altered mental status (Nervous system disorders) | 1 (1) | 0 (0)
Seizure (Nervous system disorders) | 1 (1) | 1 (1)
Thromboembolic event (Vascular disorders) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1)
Wound complication (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1/Hypermutated Phenotype (HMP) (N=8) | Cohort 2/Non-hypermutated Phenotype (NHMP). (N=30)
Abducens nerve disorder (Nervous system disorders) | 0 (0) | 1 (1)
Adrenal insufficiency (Endocrine disorders) | 0 (0) | 2 (2)
Agitation (Psychiatric disorders) | 0 (0) | 1 (1)
Alanine aminotransferase increased (Investigations) | 1 (1) | 1 (2)
Alkaline phosphatase increased (Investigations) | 0 (0) | 1 (1)
Alopecia (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Anemia (Blood and lymphatic system disorders) | 1 (1) | 1 (2)
Anorexia (Metabolism and nutrition disorders) | 0 (0) | 2 (2)
Anxiety (Psychiatric disorders) | 0 (0) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 2 (2) | 0 (0)
Ataxia (Nervous system disorders) | 2 (2) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Blood bilirubin increased (Investigations) | 0 (0) | 1 (1)
Blurred vision (Eye disorders) | 0 (0) | 1 (1)
Bronchial infection (Infections and infestations) | 1 (1) | 0 (0)
CD4 lymphocytes decreased (Investigations) | 0 (0) | 1 (1)
Cataract (Eye disorders) | 0 (0) | 1 (2)
Cognitive disturbance (Nervous system disorders) | 1 (1) | 1 (1)
Concentration impairment (Nervous system disorders) | 0 (0) | 2 (2)
Confusion (Psychiatric disorders) | 1 (2) | 2 (4)
Conjunctivitis (Infections and infestations) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 0 (0) | 2 (2)
Dizziness (Nervous system disorders) | 0 (0) | 2 (2)
Dry mouth (Gastrointestinal disorders) | 0 (0) | 1 (1)
Dysarthria (Nervous system disorders) | 0 (0) | 1 (1)
Dysesthesia (Nervous system disorders) | 1 (1) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 2 (2) | 0 (0)
Dysphasia (Nervous system disorders) | 1 (1) | 1 (1)
Eczema (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Enterocolitis infectious (Infections and infestations) | 0 (0) | 1 (1)
Eye disorders - Other, specify: decreased right peripheral vision (Eye disorders) | 0 (0) | 1 (1)
Facial muscle weakness (Nervous system disorders) | 1 (1) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 2 (3) | 2 (3)
Fatigue (General disorders) | 2 (2) | 2 (2)
Folliculitis (Infections and infestations) | 0 (0) | 1 (1)
Gait disturbance (General disorders) | 3 (4) | 5 (6)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastrointestinal disorders - Other, specify: Enteritis (Gastrointestinal disorders) | 0 (0) | 1 (2)
Gastrointestinal disorders - Other, specify: Immune-mediated colitis (Gastrointestinal disorders) | 0 (0) | 1 (2)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Hallucinations (Psychiatric disorders) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 8 (10)
Hearing impaired (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Hematuria (Renal and urinary disorders) | 0 (0) | 1 (1)
Hepatobiliary disorders - Other, specify: immune-mediated hepatitis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 0 (0) | 3 (3)
Hyperthyroidism (Endocrine disorders) | 1 (1) | 0 (0)
Hyperuricemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypocalcemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypokalemia (Metabolism and nutrition disorders) | 0 (0) | 2 (2)
Hypothyroidism (Endocrine disorders) | 1 (2) | 4 (4)
Infections and infestations - Other, specify: COVID-19 (Infections and infestations) | 1 (1) | 2 (2)
Infusion related reaction (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Insomnia (Psychiatric disorders) | 1 (1) | 0 (0)
Lethargy (Nervous system disorders) | 0 (0) | 1 (1)
Lipase increased (Investigations) | 1 (1) | 1 (2)
Lymphocyte count decreased (Investigations) | 0 (0) | 5 (10)
Memory impairment (Nervous system disorders) | 1 (1) | 1 (1)
Muscle cramp (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Muscle weakness left-sided (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2)
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Muscle weakness right-sided (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Muscle weakness upper limb (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Nausea (Gastrointestinal disorders) | 0 (0) | 5 (6)
Nervous system disorders - Other, specify: aphasia - word-finding difficulty (Nervous system disorders) | 0 (0) | 1 (1)
Nervous system disorders - Other, specify: myoclonus (Nervous system disorders) | 1 (1) | 0 (0)
Neutrophil count decreased (Investigations) | 1 (1) | 1 (3)
Pain (General disorders) | 0 (0) | 1 (1)
Pancreatitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Papulopustular rash (Infections and infestations) | 0 (0) | 2 (2)
Paresthesia (Nervous system disorders) | 0 (0) | 2 (2)
Personality change (Psychiatric disorders) | 1 (1) | 0 (0)
Platelet count decreased (Investigations) | 0 (0) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (2)
Rash acneiform (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 (0) | 4 (4)
Renal calculi (Renal and urinary disorders) | 0 (0) | 1 (1)
Seizure (Nervous system disorders) | 4 (5) | 4 (4)
Skin and subcutaneous tissue disorders - Other, specify: Right eye erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Somnolence (Nervous system disorders) | 0 (0) | 1 (1)
Surgical and medical procedures - Other, specify: Dental Root Canal (Surgical and medical procedures) | 0 (0) | 1 (1)
Thrush (Infections and infestations) | 1 (1) | 0 (0)
Upper respiratory infection (Infections and infestations) | 0 (0) | 1 (1)
Urinary incontinence (Renal and urinary disorders) | 1 (1) | 1 (1)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1) | 2 (2)
White blood cell decreased (Investigations) | 1 (1) | 1 (1)
Wound complication (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Wound infection (Infections and infestations) | 1 (1) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol and Statistical Analysis Plan (2023-03-24): https://cdn.clinicaltrials.gov/large-docs/67/NCT03718767/Prot_SAP_000.pdf
  • Informed Consent Form: Cohort Screening Consent (2023-07-26): https://cdn.clinicaltrials.gov/large-docs/67/NCT03718767/ICF_001.pdf
  • Informed Consent Form: Cohort Standard Consent (2024-11-04): https://cdn.clinicaltrials.gov/large-docs/67/NCT03718767/ICF_002.pdf